CLINICAL TRIAL: NCT04921696
Title: Association of Red Blood Cell Transfusion, Anemia, and Necrotizing Enterocolitis
Status: Withdrawn | Type: Observational
Why Stopped: no patients were included
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: NECandRBC
Record Dates: First submitted 2021-06-06; First posted 2021-06-10 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-10

CONDITIONS: Necrotizing Enterocolitis; Anemia; Red Blood Cell (RBC) Transfusion
Keywords: necrotizing enterocolitis; anemia; red blood cell (RBC) transfusion
MeSH Terms: conditions — Enterocolitis, Necrotizing; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RBC transfusion: RBC was transfused to the infants.
  Interventions: Other: RBC transfusion
- no-RBC transfusion: RBC was not transfused to the infants.
  Interventions: Other: no-RBC transfusion

INTERVENTIONS:
Other: RBC transfusion — RBC was transfused to the infants.
  Groups: RBC transfusion
Other: no-RBC transfusion — RBC was not transfused to the infants.
  Groups: no-RBC transfusion

SUMMARY:
Necrotizing enterocolitis (NEC) is a leading cause of mortality among preterm infants.The pathogenesis of NEC remains unclear with conflicting data regarding the role of red blood cell (RBC) transfusion and anemia. A meta-analysis of retrospective studies demonstrated an association between exposure to RBC transfusion and NEC(adjusted odds ratio, 2.0 [95% confidence interval, 1.6-2.5]). However, recent observational studies have found no association between RBC transfusion and NEC or have found RBC transfusion to be protective.

DETAILED DESCRIPTION:
Improving understanding of the role of RBC transfusion and anemia in the development of NEC is important. Several studies characterizing the associations between transfusion, anemia, and NEC were potentially limited by small sample size, study design. As such, researchers have underscored the need for prospective study in which each RBC exposure, episode of anemia, and outcome of NEC can be systematically and consistently evaluated.

This prospective study examined whether RBC transfusion and anemia were associated with the rate of NEC. The primary objective was to test whether NEC was increased in infants receiving RBC transfusion compared with non transfused infants. Further, exposure to severe neonatal anemia was examined as an independent risk factor for NEC.

ELIGIBILITY:
Inclusion Criteria:

* age between 1 min and 28 days
* the level blood bilirubin reached the criteria of transfusion therapy

Exclusion Criteria:

* congenital abnormalities
* receipt of transfusion before enrollment
* parents' decision not to participate
* infant not expected to survive beyond 7 days of life based on the assessment by the treating neonatologist

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The level of blood bilirubin of the included neonatal infants reached the cirteria of transfusion therapy. Whether or not the transfusion therapy was dicided according to the parents' decision.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Necrotizing enterocolitis | within 28 days
  Necrotizing enterocolitis was diagnosed within 28 days

SECONDARY OUTCOMES:
death | within 28 days
  the infant died

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China